CLINICAL TRIAL: NCT01435239
Title: The Comparison of Two Different Methods of Partial Inflation of Cuff for Facile Insertion of Laryngeal Mask Airway in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jeong-Rim LEE, Assistant Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1-2011-0046
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Surgical Complications From General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- resting volume group (Experimental)
  Interventions: Device: The cuff inflation by the resting volume
- maximum volume group (Active Comparator)
  Interventions: Device: The cuff inflation by the maximum volume

INTERVENTIONS:
Device: The cuff inflation by the resting volume — 80 patients are randomly allocated into two groups : resting volume group (n=40), half the maximum volume group (n=40). In the resting volume group, the pilot balloon valve is connected to syringe without piston for keeping the valve open to the atmosphere and allowing the pressure within the cuff of LMA to equalize with atmospheric pressure. In the half the maximum volume group, the cuff of LMA is completely emptied and then the cuff is filled with the half the maximum volume.
  Arms: resting volume group
Device: The cuff inflation by the maximum volume — 80 patients are randomly allocated into two groups : resting volume group (n=40), half the maximum volume group (n=40). In the resting volume group, the pilot balloon valve is connected to syringe without piston for keeping the valve open to the atmosphere and allowing the pressure within the cuff of LMA to equalize with atmospheric pressure. In the half the maximum volume group, the cuff of LMA is completely emptied and then the cuff is filled with the half the maximum volume.
  Arms: maximum volume group

SUMMARY:
Partial cuff inflation before insertion is generally used for laryngeal mask airway insertion in children. However, it is not proven how much the cuff should be inflated. The aim of this study is to compare efficacy between the method using the resting volume and the method using half the maximum volume for partial cuff inflation.

ELIGIBILITY:
Inclusion Criteria:

* children (0-9 years of age)
* children who is scheduled for elective surgery of short duration (less than 2 hr) undergoing general anesthesia using LMA-classic

Exclusion Criteria:

* patients with an abnormal airway
* patients with reactive airway disease
* patients with gastroesophageal reflux disease
* patients with chronic respiratory disease
* patients who has a history of an upper respiratory tract infection in the preceding 6-week period

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The intra-cuff pressure | approximately 5 to 10 minutes after insertion of LMA.
  1) After insertion of LMA, we confirm adequate ventilation. And then we measure intra-cuff pressure using cuff pressure manometer. 2) After confirming adequate ventilation, tidal volumes are measured using spirometer sensor attached anesthesia machine. Five corresponding inspiratory and expiratory tidal volumes are recorded and the difference between these is calculated as the leak volume. The time that measures the intra-cuff pressure and leak volume is approximately 5 to 10 minutes after insertion of LMA.
The leak volume | approximately 5 to 10 minutes after insertion of LMA.
  1) After insertion of LMA, we confirm adequate ventilation. And then we measure intra-cuff pressure using cuff pressure manometer. 2) After confirming adequate ventilation, tidal volumes are measured using spirometer sensor attached anesthesia machine. Five corresponding inspiratory and expiratory tidal volumes are recorded and the difference between these is calculated as the leak volume. The time that measures the intra-cuff pressure and leak volume is approximately 5 to 10 minutes after insertion of LMA.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Wallace CJ, Chambers NA, Erb TO, von Ungern-Sternberg BS. Pressure volume curves of paediatric laryngeal mask airways. Anaesthesia. 2009 May;64(5):527-31. doi: 10.1111/j.1365-2044.2008.05819.x. PMID 19413823